CLINICAL TRIAL: NCT02621905
Title: Steady-State Comparative Bioavailability Study in Patients Requiring Anti-Fungal Prophylaxis Comparing Twice a Day Dosing of Lozanoc® (Mayne) Regardless of Food With Sporanox® (Janssen) Under Fed Conditions
Brief Title: Steady-State Comparative Bioavailability Study in Prophylaxis Patients of Lozanoc® 50 mg With Sporanox® 100 mg
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Mayne Pharma International Pty Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: MPG010
Record Dates: First submitted 2015-12-02; First posted 2015-12-04 (Estimated); Last update posted 2018-10-26 (Actual); Status verified 2018-10

CONDITIONS: Neutropenia
Keywords: Prophylaxis; Steady-State; Bioavailability
MeSH Terms: conditions — Neutropenia | interventions — Itraconazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sporanox (Active Comparator): 100 mg
  Interventions: Drug: Sporanox
- Lozanoc (Experimental): 50 mg
  Interventions: Drug: Lozanoc

INTERVENTIONS:
Drug: Sporanox — At least 2 capsules twice a day for 3 weeks
  Other Names: itraconazole
  Arms: Sporanox
Drug: Lozanoc — At least 2 capsules twice a day for 3 weeks
  Other Names: itraconazole
  Arms: Lozanoc

SUMMARY:
The pharmacokinetics of Sporanox and Lozanoc has not been compared in patients requiring anti-fungal prophylaxis or therapy. The present study is designed to compare the pharmacokinetics of Sporanox and Lozanoc in patients requiring primary prophylaxis. The 3-week exposure to each formulation is designed to allow for all participants to reach steady-state for each drug, as the time to steady-state can vary.

DETAILED DESCRIPTION:
After confirmation of eligibility, participants will be randomly assigned 1:1 to commence therapy with either 100mg mane and 100mg nocte for 21 days or Sporanox 200mg mane and 200mg nocte with food for 21 days. If a subject enters the study already receiving itraconazole prophylaxis at a dose of itraconazole higher than 100 mg twice a day, the subject will then be dosed on study at the pre-study dosage; that is, the subject will take the same number of capsules per day on study as the subject was taking prior to enrolment in the study.

The following information will be collected at baseline; whether the participant is taking itraconazole prophylaxis and at what dose; whether the participant is taking gastric suppression therapy. Patients who are not taking food or who are taking gastric acid suppression therapy (antacids, an H2 antagonist or a proton pump inhibitor) can take Sporanox with cola or orange juice to maximise absorption as recommended in the Sporanox product label (not required for Lozanoc formulation).

At Day 22, participants assigned to

* Lozanoc and who have completed 21 days of Lozanoc prophylaxis will cross over to the same number of Sporanox capsules with food for a further 21 days
* Sporanox and who have completed 21 days of Sporanox prophylaxis will cross over to the same number of Lozanoc capsules for a further 21 days.

The dose of either drug may be dose-reduced or ceased for toxicity at the discretion of the investigator.

During the course of the treatment periods participants will undergo the following assessments:

* Concurrent medication(s)
* Clinical adverse events
* Measurement of vital signs (weight, blood pressure, temperature)
* Targeted physical examination
* Documentation of any evidence of systemic fungal infection
* Medication and meal diaries
* 12-lead electrocardiogram (ECG)
* Laboratory safety assessments: Renal function and electrolytes (urea, creatinine, estimated glomerular filtration rate [eGFR], sodium, potassium, chloride, bicarbonate), Liver function tests (bilirubin, albumin, total protein, alanine aminotransferase [ALT], aspartate aminotransferase [AST])
* Pharmacokinetic testing: Trough (pre-morning dose; 0 hr) sample will be collected at Baseline (Day 1), and at Days 8, 15, 22, 29, 36 and 43. Post-dose samples will also be collected 2, 3.5 and 6 hours after the morning dose on Day 22 and Day 43

ELIGIBILITY:
Inclusion Criteria:

* Provision of written, informed consent
* Age of at least 18 years
* No clinical evidence of active systemic fungal infection
* Physician-recommended primary prophylaxis against systemic fungal infections with itraconazole in patients who have had or about to have: a heart, lung or bone marrow transplant, combination chemotherapy for cancer; aspergilloma, chronic pulmonary aspergillus bronchitis, or allergic bronchopulmonary aspergillosis
* Patients may be receiving itraconazole prophylaxis prior to entry into the study
* Body mass index between 15.0 and 35.0 kg/m2

Exclusion Criteria:

* Pregnant, planning pregnancy or breastfeeding
* Congestive cardiac failure or other causes of ventricular dysfunction that may outweigh the benefit of itraconazole
* Hypersensitivity to either study drug or to any of their excipients
* Coadministration of the following drugs:

  * CYP3A4 metabolised substrates that can prolong the QT-interval e.g., sertindole, terfenadine
  * CYP3A4 metabolised HMG-CoA reductase inhibitors e.g. simvastatin, lovastatin
  * Potent CYP3A4 inhibitors e.g. dronedarone
  * Triazolam, alprazolam and oral midazolam
  * Ergot alkaloids such as dihydroergotamine, ergometrine (ergonovine) and ergotamine

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2015-11 (Actual); Primary Completion 2016-11 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Relative steady-state bioavailability | 3 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Deborah Marriott, Principal Investigator — St Vincent's Hospital, Sydney
Locations (1):
- St Vincent's Hospital, Darlinghurst, New South Wales, Australia

IPD SHARING:
Plan to Share IPD: No
Individual patient data will not be made available